CLINICAL TRIAL: NCT03608306
Title: Clinical Performance of Bioactive Restorative Material Versus Glass Hybrid Restorative in Posterior Restorations of High Caries Risk Patients: Randomized Clinical Trial
Brief Title: Clinical Performance of Bioactive Restorative Material Versus Glass Hybrid Restorative in Posterior Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona mahmoud Abd Elrahman, Principal Investigator and PHD student at Conservative Dentistry Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-07-11
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Dental Restoration Failure
Keywords: Clinical Performance; Bioactive Restorative Material; Glass Hybrid Restorative
MeSH Terms: interventions — ACTIVA BioACTIVE-RESTORATIVE

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin-modified glass ionomer (Experimental): Activa Bioactive-Restorative is an enhanced resin modified glass ionomer (RMGI) with an ionic resin matrix, a shock-absorbing resin component, and bioactive fillers that mimic the physical and chemical properties of natural teeth.
  Interventions: Other: Resin-modified glass ionomer
- Bulk-fill glass hybrid restorative (Active Comparator): EQUIA Forte is a bulk-fill, fluoride-releasing restorative system that combines EQUIA Forte Fil, which is a high strength glass hybrid restorative, and EQUIA Forte Coat, a wear-resistant, self-adhesive, light-cured resin coating.
  Interventions: Other: Bulk-fill glass hybrid restorative

INTERVENTIONS:
Other: Resin-modified glass ionomer — enhanced RMGIs with an ionic resin matrix, a shock-absorbing resin component, and bioactive fillers that mimic the physical and chemical properties of natural teeth.
  Other Names: Activa Bioactive-Restorative
  Arms: Resin-modified glass ionomer
Other: Bulk-fill glass hybrid restorative — It's a bulk-fill, fluoride-releasing restorative system that combines EQUIA Forte Fil, which is a high strength glass hybrid restorative, and EQUIA Forte Coat, a wear-resistant, self-adhesive, light-cured resin coating.
  Other Names: EQUIA Forte
  Arms: Bulk-fill glass hybrid restorative

SUMMARY:
Clinical performance of bioactive restorative material versus glass hybrid restorative in posterior restorations of high caries risk patients will be evaluated over 12 months using Fédération Dentaire Internationale' (FDI) clinical criteria for the evaluation of direct and indirect restorations

DETAILED DESCRIPTION:
The application of resin composite has been described as "technique sensitive". Although glass ionomers are inferior to resin composite in esthetics, there are specific clinical situations where glass ionomers are the materials of choice for restoring teeth as patients at risk for caries and with carious lesions due to its ability to release fluoride and to self-adhere to enamel and dentin.

However, Conventional glass ionomer have poor physical and mechanical properties and are more liable to wear when compared to resin composite. The change in formulation of resin modified glass ionomer restorations allowed them to have improved physic-mechanical properties, combined with significant improvement in esthetic properties. Thus, in recent years glass ionomer as direct restorative materials have become more user friendly. Unfortunately, most of glass ionomers are not recommended as definitive final restorations for the permanent dentition in stress bearing areas because they do not have the physical and mechanical properties of amalgam or composite resin.

ACTIVA™ BioACTIVE-RESTORATIVE™ is recently introduced enhanced resin modified glass ionomer, which the manufacturer (Pulpdent Corporation, USA) reports to be the first bioactive dental materials with an ionic resin matrix, a shock-absorbing resin component, and bioactive fillers that mimic physical and chemical properties of natural teeth. They are durable, fracture and wear resistant, chemically bond to teeth, seal against bacterial microleakage, and release and recharge with calcium, phosphate, and more fluoride ions than glass ionomers. Thus, ACTIVA has more release and recharge of calcium, phosphate and fluoride than glass ionomers with the esthetics, strength, and physical properties of composites, combining the best attributes of both materials without compromising either one.

EQUIA® Forte is a fluoride-releasing, bulk-fill system which consists of EQUIA® Forte Fil, a high strength glass hybrid restorative, and EQUIA® Forte Coat, a wear-resistant, self-adhesive, light-cured resin coating. With improved flexural strength, and acid and wear resistance, the manufacturer claims that EQUIA® Forte extends the recommended indications to include stress-bearing Class II restorations.

The clinical performance of these materials regarding functional, esthetic and biological properties is yet to be evaluated. The FDI clinical criteria provide more detailed evaluation criteria and better differentiation between different types of failure; and incorporate objective assessment tools and a clear scoring system than other scoring systems. Thus, this study aims to contribute to providing evidence-based literature concerning current innovative Resin-modified glass ionomer restorations using the most updated and standardized assessment criteria, namely the FDI.

ELIGIBILITY:
Inclusion Criteria:

* High caries risk patients with multiple posterior cavitated carious lesions
* Co-operative patients approving to participate in the study.
* Pulp asymptomatic vital carious posterior teeth.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Low caries risk patients.
* Anterior carious lesions
* Lack of compliance
* Severe medical complications.
* Pregnancy.
* Evidence of parafunctional habits
* Temporomandibular joint disorders
* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in the clinical performance using Fédération Dentaire Internationale' (FDI) World Dental Federation clinical criteria for the evaluation of direct and indirect restorations | Change from the baseline at 6 months and12 months
  (FDI) criteria includes :
  * Biological properties (Postoperative hypersensitivity & tooth vitality, Recurrence of caries, erosion & abfraction,Tooth integrity (enamel cracks or tooth fractures),Periodontal response (compared to a reference tooth),Adjacent mucosa, Oral & general health)
  * Esthetic properties (Surface luster, Staining (surface &margin),Color match & translucency & Esthetic anatomical form)
  * Functional properties (Fracture or material retention, Marginal integrity, Occlusal contour &wear (quantitatively & qualitatively), Proximal anatomical form(contact point &contour), Radiographic examination(when applicable) &Patient's view)
  For each criteria one score will be chosen from 5 scores (excellent, good, satisfactory, unsatisfactory & poor).
  Subscales will not be combined

CONTACTS AND LOCATIONS:
Overall Officials: Mai M Yousry, PhD, Study Director — Professor of Conservative Dentistry, Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bansal R, Burgess J, Lawson NC. Wear of an enhanced resin-modified glass-ionomer restorative material. Am J Dent. 2016 Jun;29(3):171-4. PMID 27505995
- [Background] Fleming GJ, Awan M, Cooper PR, Sloan AJ. The potential of a resin-composite to be cured to a 4mm depth. Dent Mater. 2008 Apr;24(4):522-9. doi: 10.1016/j.dental.2007.05.016. Epub 2007 Jul 31. PMID 17669481
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Clin Oral Investig. 2007 Mar;11(1):5-33. doi: 10.1007/s00784-006-0095-7. Epub 2007 Jan 30. PMID 17262225
- [Background] Pameijer CH, Garcia-Godoy F, Morrow BR, Jefferies SR. Flexural strength and flexural fatigue properties of resin-modified glass ionomers. J Clin Dent. 2015;26(1):23-7. PMID 26054188